CLINICAL TRIAL: NCT02201472
Title: Magnetic Resonance Elastography in Infants
Acronym: MREI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of research focus
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-3065
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2017-02

CONDITIONS: Liver Disease
Keywords: liver; mre; mri; neonatal; mr touch
MeSH Terms: conditions — Liver Diseases | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: Magnetic resonance elastography on infants with suspected liver disease
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI with MRE (Experimental): Magnetic Resonance Imaging with Magnetic Resonance Elastography using the GE MR Touch device
  Interventions: Device: MRI with MRE

INTERVENTIONS:
Device: MRI with MRE — Magnetic Resonance Imaging with Magnetic Resonance Elastography using the GE MR Touch device

SUMMARY:
MRI & MRE in infants

DETAILED DESCRIPTION:
The purpose of the present pilot study is to determine the feasibility of using MRI and MRE to evaluate the liver in infants with suspected liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 6 months of age
* Known liver disease based (liver enzymes, bilirubin, and/or GGT at least twice the upper limit of normal for age)
* Parental/LAR permission obtained

Exclusion Criteria:

* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology
* Severe coagulopathy (INR > 3 or platelets <50,000)

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Merhar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI With MRE
Started | 2
Completed | 0
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Study closed due to low enrollment. The two participants that were enrolled did not have their data analyzed.
Arm/Group | MRI With MRE
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: months]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of MRE to Provide Evaluable Images That Illustrate the Stiffness of Liver Parenchyma in an Infant Population
Description: To determine the feasibility of MRE to provide evaluable images that illustrate the stiffness of liver parenchyma in an infant population.
Time Frame: 12 months
Population: There were too few eligible candidates that clinically would benefit enough to justify the potential risk of being removed from the unit and undergoing MRE in a Radiology department scanner, so the study was terminated with only 2 patients enrolled.
Arm/Group | MRI With MRE
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MRI With MRE
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Due to difficulty with finding neonates who met the inclusion/exclusion criteria who were safe to leave the NICU and go to the Radiology department, the study was terminated and data from the 2 participants enrolled was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes